CLINICAL TRIAL: NCT00000632
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of 100 mcg of Env 2-3 in MF59
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Biocine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Prevention
Other Study IDs: AVEG 005C; 10548 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Vaccines, Synthetic; Drug Evaluation; Adjuvants, Immunologic; AIDS Vaccines; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: Env 2-3

SUMMARY:
To evaluate the safety and immune response of 100 mcg Env 2-3 antigen administered on days 0, 30, 180, and 365.

Preliminary immunologic data from protocol VEU 005B show evidence of the development of functional antibodies in the form of increased peptide binding and development of neutralizing antibodies. Evaluation of an antigen dose having potentially greater immunogenicity is therefore of particular interest.

DETAILED DESCRIPTION:
Preliminary immunologic data from protocol VEU 005B show evidence of the development of functional antibodies in the form of increased peptide binding and development of neutralizing antibodies. Evaluation of an antigen dose having potentially greater immunogenicity is therefore of particular interest.

Twelve healthy volunteers receive injections of 100 mcg Env 2-3 in MF59 emulsion and two volunteers receive MF59 only on days 0, 30, 180, and 365. Follow-up continues for 6 months after the last injection.

ELIGIBILITY:
Inclusion Criteria

Subjects are:

* Normal, healthy adults (by history and physical examination) who fully comprehend the purpose and details of the study.

Exclusion Criteria

Co-existing Condition:

Subjects with the following conditions or symptoms are excluded:

* Positive syphilis serology (such as VDRL) unless positive test is due to a documented clinical event that occurred and was treated 5 or more years prior to enrollment.
* Circulating hepatitis B antigenemia.

Subjects with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, or autoimmune disease.
* Evidence of depression or under treatment for psychiatric problems during the past year.

Prior Medication:

Excluded:

* Immunosuppressive medications.

Prior Treatment:

Excluded:

* Blood transfusions or cryoprecipitates within the past 6 months.

Identifiable high-risk behavior for HIV infection, including:

* history of intravenous drug use; syphilis, gonorrhea, or any other sexually transmitted diseases (including chlamydia or pelvic inflammatory disease) in the last 6 months; more than two sexual partners, or sexual contact with a high-risk partner, in the preceding 6 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Study Completion 1992-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dolin R, Study Chair
Locations (3):
- United States (3):
  - Univ. of Rochester AVEG, Rochester, New York
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee
  - UW - Seattle AVEG, Seattle, Washington

REFERENCES:
- [Background] Evans TG, Fitzgerald T, Gibbons DC, Keefer MC, Soucier H. Th1/Th2 cytokine responses following HIV-1 immunization in seronegative volunteers. The AIDS Vaccine Evaluation Group. Clin Exp Immunol. 1998 Feb;111(2):243-50. doi: 10.1046/j.1365-2249.1998.00486.x. PMID 9486388
- [Background] Keefer MC, Graham BS, McElrath MJ, Matthews TJ, Stablein DM, Corey L, Wright PF, Lawrence D, Fast PE, Weinhold K, Hsieh RH, Chernoff D, Dekker C, Dolin R. Safety and immunogenicity of Env 2-3, a human immunodeficiency virus type 1 candidate vaccine, in combination with a novel adjuvant, MTP-PE/MF59. NIAID AIDS Vaccine Evaluation Group. AIDS Res Hum Retroviruses. 1996 May 20;12(8):683-93. doi: 10.1089/aid.1996.12.683. PMID 8744579